CLINICAL TRIAL: NCT02224456
Title: A Prospective, Multi-center, Cohort Study to Evaluate the Efficacy and Safety of Tenofovir Disoproxil Fumarate (TDF) Therapy in Chinese Chronic Hepatitis B (CHB) Subjects With Advanced Fibrosis & Compensated Cirrhosis
Brief Title: Efficacy and Safety Study of Tenofovir Disoproxil Fumarate (TDF) in Chinese Chronic Hepatitis B (CHB) Subjects With Advanced Fibrosis & Compensated Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201213
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-11

CONDITIONS: Hepatitis B, Chronic
Keywords: Tenofovir disoproxil fumarate; hepatocellular carcinoma; chronic hepatitis B; Cirrhosis
MeSH Terms: conditions — Hepatitis B, Chronic; Carcinoma, Hepatocellular; Fibrosis | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tenofovir (Experimental): Subjects will receive TDF 300 milligrams (mg) tablet once daily for 240 weeks in the study. Subjects who receive add-on rescue treatment may take LAM 100 mg, ETV 0.5 mg or LdT 600 mg per day upon investigator's decision in addition to TDF tablet.
  Interventions: Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — White, almond-shaped, film-coated tablet containing 300 mg of TDF, debossed with "GILEAD" and "4331" on one side of the tablet.

SUMMARY:
Chronic Hepatitis B infection (CHB) is known as the most frequently identified cause of liver disease that predisposes patients to the development of hepatocellular carcinoma (HCC). Active hepatitis B virus (HBV) replication is the key driver of liver injury and disease progression. Majority of Chinese patients are infected with genotype B and C HBV, which is different from Caucasian counterparts. This prospective multi-center cohort open-label study is designed to investigate the long-term effect of TDF on prevention of HCC and disease progression as well as to evaluate the efficacy and safety of long-term TDF in Chinese CHB subjects with advanced liver diseases. The study will enrol 240 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years(inclusive);
* Presence of HBsAg in serum at screening and for at least 6 months before screening assessment;
* Serum HBV DNA>=2000 IU/mL if HBeAg positive at screening (with or without ALT elevation); or serum HBV DNA>=200IU/mL if HBeAg negative at screening (with or without ALT elevation);
* Clinically diagnosed as advanced fibrosis or compensated cirrhosis defined as both of following : liver stiffness measure (LSM) >12.4 kiloPascals (kpa) (ALT> Upper limit of normal [ULN]) or LSM>9.0 kpa (ALT<=ULN); One of following: Liver biopsy showing advanced fibrosis or cirrhosis (Ishak score >=4, within the previous 6 months before screening and provided that no treatment likely to improve liver histology has been taken since). The slides must be available for review by an independent histopathologist; Endoscopy-proven gastroesophageal or gastric varices, non-cirrhotic portal hypertension excluded; Abdominal ultrasound or CT found changes indicating cirrhosis, irregular liver surface or nodularity, with/without splenomegaly (depth of spleen>4.0cm or spleen length>13cm); Blood platelets <100 x10^9/L (and other causes of thrombocytopenia excluded);
* Ability to give written informed consent;
* A female is eligible to enter and participate in this study if she is of: non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal), or Child-bearing potential, has a negative urine pregnancy test at screening, and agrees to one of the following methods for avoidance of pregnancy during the period of the study and until 30 days after last dose of study medication: Oral contraceptive, either combined or progestogen alone; Injectable progestogen; Implants of levonorgestrel; Oestrogenic vaginal ring; Percutaneous contraceptive patches; Intrauterine device (IUD) or intrauterine system (IUS) showing that the expected failure rate is less than 1% per year as stated in the IUD or IUS product label; Has a male partner who is sterilised; Double barrier method: condom and an occlusive cap (diaphragm orcervical/vault caps) with a vaginal spermicidal agent (foam/gel/film /cream/suppository).
* Agreement not to participate in any other investigational trials or to undertake other HBV systemic antiviral or interferon (IFN) regimens during participation in this study.

Exclusion Criteria:

* Hepatocellular carcinoma as evidenced by one of the following: Suspicious foci on ultrasound or radiological examination; Normal ultrasound serum alpha-fetoprotein >50 nanograms (ng)/mL at screening.
* Serum ALT >10 times ULN at screening or history of acute exacerbation leading to transient decompensation;
* Documented co-infection with hepatitis A (HAV), hepatitis C (HCV), hepatitis delta virus (HDV), hepatitis E virus (HEV) or human immunodeficiency virus (HIV). For HCV co-infection, subjects who are anti-HCV positive and in whom HCV ribonucleic acid (RNA) is undetectable are considered to be not eligible for enrolment.
* Evidence of active liver disease due to autoimmune hepatitis (antinuclear antibody (ANA) titre >1:160).
* Decompensated liver disease as indicated by any of the following: serum bilirubin >1.5 xULN prothrombin time activity <60% or International normalized ratio (INR)>1.5; serum albumin <32 grams per liter (g/L); history of previous clinical hepatic decompensation (e.g., ascites, variceal bleeding, or encephalopathy);
* Planned for liver transplantation or previous liver transplantation;
* Creatinine clearance less than 70 mL/minute (min);
* Haemoglobin <10 g/deciliter (dL), white blood cell (WBC) count <1.5 x 10^9/liter (L), platelets <=50 x 10^9/L;
* Any serious or active medical or psychiatric illnesses other than hepatitis B which, in the opinion of the Investigator, would interfere with subject treatment, assessment or compliance with the protocol. This would include any uncontrolled clinically significant renal, cardiac, pulmonary, vascular, neurogenic, digestive, metabolic (diabetes, thyroid disorders, adrenal disease), immunodeficiency disorders, pathological fractures or cancer;
* Active alcohol or drug abuse or history of alcohol or drug abuse considered by the Investigator to be sufficient to hinder compliance with treatment, participation in the study or interpretation of results;
* A female who is breastfeeding or plan to breastfeed;
* Use of immunosuppressive therapy, immunomodulatory therapy (including IFN or thymosin alpha), systemic cytotoxic agents, chronic antiviral agents including Chinese herbal medicines known to have activity against HBV (e.g., lamivudine (LAM), adefovir, entecavir (ETV), telbivudine (LdT) or hepatitis B immunoglobulin (HBIg)) within the previous 6 months prior to screening into this study;
* Have ever received TDF or any medicinal products containing the above mentioned antiviral agents or any investigative anti-HBV treatments (e.g., emtricitabine (FTC), (2R,4R)-4-(2,6-Diaminopurin-9-yl)-1,3-dioxolan-2-yl]methanol (DAPD) and 1-(2-fluoro-5-methyl-beta, Larabinofuranosyl) uracil (L-FMAU));
* History of hypersensitivity to nucleoside and/or nucleotide analogues and/or any component of study medication;
* Therapy with nephrotoxic drugs (e.g., aminoglycosides, amphotercin B, vancomycin, cidofovir, foscarnet, cis-platinum, pentamidine etc.) or competitors of renal excretion (e.g., probenecid) within 2 months prior to study screening or the expectation that subject will receive any of these during the course of the study;
* Inability to comply with study requirements as determined by the study Investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- China (14):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Xian, Shanxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Taiyuan
  - GSK Investigational Site, Xi'an
  - GSK Investigational Site, Zhengzhou

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted to evaluate the efficacy and safety of 300 milligram (mg) Tenofovir Disoproxil Fumarate (TDF) therapy in Chinese chronic hepatitis B (CHB) participants with advanced fibrosis and compensated cirrhosis
Pre-assignment Details: A total of 266 participants were screened, of which 197 entered the study.
Groups:
- Tenofovir Disoproxil Fumarate 300 mg: Participants received Tenofovir Disoproxil Fumarate 300 mg tablet once daily (QD) orally for 240 weeks.
Period: Overall Study
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Started | 197
Completed | 161
Not Completed | 36
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 15
Not completed — Withdrawal by Subject | 9
Not completed — Physician Decision | 3
Not completed — Death | 2
Not completed — Pregnancy | 4
Not completed — Protocol Violation | 1
Not completed — Treatment Interruptions of ≥28 days | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics is presented for modified Intent-to-treat (mITT) Population which consisted of all participants who received at least one dose of study medication. 2 participants did not receive TDF treatment thus excluded from mITT Population
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics is presented for mITT Population which consisted of all participants who received at least one dose of study medication. 2 participants did not receive TDF treatment thus excluded from mITT Population
  Years | 42.3 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics is presented for mITT Population which consisted of all participants who received at least one dose of study medication. 2 participants did not receive TDF treatment thus excluded from mITT Population
  Participants
    Female | 47
    Male | 148
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Baseline characteristics is presented for mITT Population which consisted of all participants who received at least one dose of study medication. 2 participants did not receive TDF treatment thus excluded from mITT Population
  Participants
    Asian | 195

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Newly Diagnosed Hepatocellular Carcinoma (HCC) at Week 240
Description: The newly diagnosed HCC was defined as HCC cases from Week 24 to Week 240 and the participants were required to meet one of the following criteria: without HCC before Week 24; a histological diagnosis of HCC (i.e. by biopsy or at post-mortem); participants with nodules >2 centimeter (cm), identification of typical HCC characteristics (hyper-vascular in the arterial phase with washout in the portal venous or delayed phases) by 4-phase multi-detector computed tomography (CT) scan or dynamic contrast-enhanced magnetic resonance imaging (MRI); participants with nodules >1 cm, identification of typical HCC characteristics by both techniques (4-phase multi-detector CT and dynamic contrast-enhanced MRI).
Time Frame: Week 240
Population: Modified Intent-to-treat (mITT) Population consisted of all recruited participants who received at least one dose of study medication.
Measure: Number; unit: Events per person-year
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 195
Events per person-year | 6.045

2. Primary Outcome: Percentage of Participants With Disease Progression at Week 240
Description: Disease progression was defined as the first occurrence of any one of the following criteria: 1) an increase in Childs-Pugh score of 2 or more points from Baseline; 2) an increase in Childs-Pugh score of 2 or more points, solely based on laboratory parameters (i.e. bilirubin, prothrombin time and/or albumin) confirmed between two consecutive visits at least one month apart; 3) spontaneous bacterial peritonitis (with proven sepsis); 4) renal insufficiency; 5) bleeding gastric/esophageal varices; 6) hepatocellular carcinoma; 7)liver-related death.
Time Frame: Week 240
Population: mITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 195
Percentage of participants | 7.2

3. Secondary Outcome: Number of Participants With Newly Diagnosed Hepatocellular Carcinoma (HCC) at Week 48, Week 96, Week 144 and Week 192
Description: as for outcome 1
Time Frame: Week 48, Week 96, Week 144 and Week 192
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 195
Participants
  Week 48 | 0
  Week 96 | 0
  Week 144 | 4
  Week 192 | 9

4. Secondary Outcome: Percentage of Participants With Newly Diagnosed Hepatocellular Carcinoma (HCC) at Week 48, Week 96, Week 144, Week 192 and Week 240
Description: The newly diagnosed HCC was defined as HCC cases from Week 24 to Week 240 and the participants were required to meet one of the following criteria: without HCC before Week 24; a histological diagnosis of HCC (i.e. by biopsy or at post-mortem); participants with nodules >2 centimeter (cm), identification of typical HCC characteristics (hyper-vascular in the arterial phase with washout in the portal venous or delayed phases) by 4-phase multi-detector computed tomography (CT) scan or dynamic contrast-enhanced magnetic resonance imaging (MRI); participants with nodules >1 cm, identification of typical HCC characteristics by both techniques (4-phase multi-detector CT and dynamic contrast-enhanced MRI).The cumulative percentage of participants with newly diagnosed Hepatocellular Carcinoma has been presented along with 95% confidence interval (CI) (Wald method).
Time Frame: Week 48, Week 96, Week 144, Week 192 and Week 240
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 195
Percentage of participants
  Week 48 | 0 [NA to NA] — NA indicates that 95% CI could not be calculated due to insufficient participants with events
  Week 96 | 0 [NA to NA] — NA indicates that 95% CI could not be calculated due to insufficient participants with events
  Week 144 | 2.1 [0.0 to 4.3]
  Week 192 | 4.6 [1.4 to 7.8]
  Week 240 | 5.6 [2.1 to 9.1]

5. Secondary Outcome: Percentage of Participants With Disease Progression at Week 48, Week 96, Week 144, Week 192 and Week 240
Description: Disease progression was defined as the first occurrence of any one of the following criteria: 1) an increase in Childs-Pugh score of 2 or more points from Baseline; 2) an increase in Childs-Pugh score of 2 or more points, solely based on laboratory parameters (i.e. bilirubin, prothrombin time and/or albumin) confirmed between two consecutive visits at least one month apart; 3) spontaneous bacterial peritonitis (with proven sepsis); 4) renal insufficiency; 5) bleeding gastric/oesophageal varices; 6) hepatocellular carcinoma; 7) liver-related death. The cumulative percentage of participants with disease progression has been presented along with 95% CI (Wald method).
Time Frame: Week 48, Week 96, Week 144, Week 192 and Week 240
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 195
Percentage of participants
  Week 48 | 2.1 [0.0 to 4.3]
  Week 96 | 2.6 [0.1 to 5.0]
  Week 144 | 4.1 [1.1 to 7.1]
  Week 192 | 7.2 [3.3 to 11.1]
  Week 240 | 7.2 [3.3 to 11.1]

6. Secondary Outcome: Mean Change From Baseline in Liver Stiffness Measure at Week 48, Week 96, Week 144, Week 192 and Week 240
Description: Liver stiffness measure was obtained by a non-invasive transient elastography using FibroScan. Baseline is defined as the last assessment (Day 0) before administration of the study drug. Change from Baseline is defined as post-dose visit value minus Baseline value
Time Frame: Baseline (Day 0), Week 48, Week 96, Week 144, Week 192 and Week 240
Population: mITT Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles.
Measure: Mean (Standard Deviation); unit: Kilopascals
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 182
Kilopascals
  Week 48, n=182 | -3.3 (4.84)
  Week 96, n= 176: number analyzed (Participants) | 176
  Week 96, n= 176 | -4.7 (5.60)
  Week 144, n= 175: number analyzed (Participants) | 175
  Week 144, n= 175 | -5.1 (5.85)
  Week 192, n=167: number analyzed (Participants) | 167
  Week 192, n=167 | -5.1 (7.82)
  Week 240, n= 131: number analyzed (Participants) | 131
  Week 240, n= 131 | -6.2 (5.55)

7. Secondary Outcome: Percentage of Participants With Serum Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) <20 International Units Per Milliliter (IU/mL) at Weeks 48, 96, 144, 192 and 240
Description: Serum samples were collected for the analysis of HBV DNA levels using Roche Cobas Taqman HBV test. Confidence interval was calculated by normal approximation and continuity correction method.
Time Frame: Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 191
Percentage of participants
  Week 48, n=191 | 81.2 [75.3 to 87.0]
  Week 96, n=188: number analyzed (Participants) | 188
  Week 96, n=188 | 88.8 [84.1 to 93.6]
  Week 144, n=185: number analyzed (Participants) | 185
  Week 144, n=185 | 94.1 [90.4 to 97.7]
  Week 192, n=174: number analyzed (Participants) | 174
  Week 192, n=174 | 97.7 [95.2 to 100.0]
  Week 240, n=160: number analyzed (Participants) | 160
  Week 240, n=160 | 99.4 [97.8 to 100.0]

8. Secondary Outcome: Change From Baseline in Logarithm to the Base 10 (Log 10) Serum HBV DNA
Description: Serum samples were collected for the analysis of HBV DNA levels. Baseline is defined as the last assessment (Day 0) before administration of the study drug. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Log 10 (IU/mL)
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 191
Log 10 (IU/mL)
  Week 48, n=191 | -4.2 (1.40)
  Week 96, n=188: number analyzed (Participants) | 188
  Week 96, n=188 | -4.3 (1.44)
  Week 144, n=185: number analyzed (Participants) | 185
  Week 144, n=185 | -4.3 (1.48)
  Week 192, n=174: number analyzed (Participants) | 174
  Week 192, n=174 | -4.2 (1.50)
  Week 240, n=160: number analyzed (Participants) | 160
  Week 240, n=160 | -4.3 (1.46)

9. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization at Week 48, Week 96, Week 144, Week 192 and Week 240 in Participants Who Had Abnormal ALT at Baseline
Description: Blood samples were collected for evaluation of ALT at indicated time points. ALT normalization is defined as ALT outside the normal range at Baseline and within the normal range at Week 48, Week 96, Week 144, Week 192 and Week 240. Normal range of ALT is 7 to 56 International Units per liter. Percentage of participants with ALT normalization at Weeks 48, 96, 144, 192 and 240 in participants who had abnormal ALT at Baseline (Day 0) have been presented. Confidence interval was calculated using normal approximation and continuity correction method.
Time Frame: Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 97
Percentage of participants
  Week 48, n=97 | 63.9 [53.8 to 74.0]
  Week 96, n= 97 | 66.0 [56.0 to 75.9]
  Week 144, n=96: number analyzed (Participants) | 96
  Week 144, n=96 | 70.8 [61.2 to 80.4]
  Week 192, n=93: number analyzed (Participants) | 93
  Week 192, n=93 | 82.8 [74.6 to 91.0]
  Week 240, n=87: number analyzed (Participants) | 87
  Week 240, n=87 | 82.8 [74.2 to 91.3]

10. Secondary Outcome: Percentage of Hepatitis B e Antigen (HBeAg) Positive Participants Achieving HBeAg Loss, HBeAg Seroconversion at Week 48, Week 96, Week 144, Week 192 and Week 240.
Description: Serological response was assessed at Week 48, Week 96, Week 144, Week 192 and Week 240 in participants with Positive HBeAg at Baseline (Day 0). It was presented as HBeAg Loss and HBeAg Seroconversion. HBeAg Loss was defined as HBeAg changed to be negative. HBeAg seroconversion was defined as HBeAg changed to negative and HBeAb was positive. Confidence interval was calculated using normal approximation and continuity correction method.
Time Frame: Week 48, Week 96, Week 144, Week 192 and Week 240
Population: mITT Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles.)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 94
Percentage of participants
  Week 48, HBeAg Loss, n=94 | 18.1 [9.8 to 26.4]
  Week 48, HBeAg Seroconversion, n=94 | 9.6 [3.1 to 16.1]
  Week 96, HBeAg , n=94 | 33.0 [22.9 to 43.0]
  Week 96, HBeAg Seroconversion, n=94 | 14.9 [7.2 to 22.6]
  Week 144, HBeAg Loss, n=90: number analyzed (Participants) | 90
  Week 144, HBeAg Loss, n=90 | 35.6 [24.5 to 45.1]
  Week 144, HBeAg Seroconversion, n=90: number analyzed (Participants) | 90
  Week 144, HBeAg Seroconversion, n=90 | 14.4 [6.5 to 21.8]
  Week 192, HBeAg Loss, n=90: number analyzed (Participants) | 90
  Week 192, HBeAg Loss, n=90 | 47.8 [36.4 to 58.1]
  Week 192, HBeAg Seroconversion, n=90: number analyzed (Participants) | 90
  Week 192, HBeAg Seroconversion, n=90 | 16.7 [8.3 to 24.7]
  Week 240, HBeAg Loss, n=82: number analyzed (Participants) | 82
  Week 240, HBeAg Loss, n=82 | 51.2 [38.7 to 61.3]
  Week 240, HBeAg Seroconversion, n=82: number analyzed (Participants) | 82
  Week 240, HBeAg Seroconversion, n=82 | 23.2 [13.1 to 32.2]

11. Secondary Outcome: Percentage of HBeAg Negative Participants Achieving HBsAg Loss and HBsAg Seroconversion at Week 48, Week 96, Week 144, Week 192 and Week 240
Description: Serological response was assessed at Week 48, Week 96, Week 144, Week 192 and Week 240 in participants with negative HBeAg at Baseline (Day 0). HBsAg Loss was defined as HBsAg changed to be negative. HBsAg seroconversion was defined as HBsAg changed to negative and HBsAb was positive.
Time Frame: Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 97
Percentage of Participants
  Week 48, HBsAg Loss, n=97 | 1.0 [0.0 to 3.6]
  Week 48, HBsAg Seroconversion, n=97 | 1.0 [0.0 to 3.6]
  Week 96, HBsAg , n=93: number analyzed (Participants) | 93
  Week 96, HBsAg , n=93 | 0 [0.0 to 0.5]
  Week 96, HBsAg Seroconversion, n=93: number analyzed (Participants) | 93
  Week 96, HBsAg Seroconversion, n=93 | 0 [0.0 to 0.5]
  Week 144, HBsAg Loss, n=93: number analyzed (Participants) | 93
  Week 144, HBsAg Loss, n=93 | 3.2 [0.0 to 7.4]
  Week 144, HBsAg Seroconversion, n=93: number analyzed (Participants) | 93
  Week 144, HBsAg Seroconversion, n=93 | 0 [0.0 to 0.5]
  Week 192, HBsAg Loss, n=89: number analyzed (Participants) | 89
  Week 192, HBsAg Loss, n=89 | 4.5 [0.0 to 9.4]
  Week 192, HBsAg Seroconversion, n=89: number analyzed (Participants) | 89
  Week 192, HBsAg Seroconversion, n=89 | 2.2 [0.0 to 5.9]
  Week 240, HBsAg Loss, n=77: number analyzed (Participants) | 77
  Week 240, HBsAg Loss, n=77 | 5.2 [0.0 to 10.8]
  Week 240, HBsAg Seroconversion, n=77: number analyzed (Participants) | 77
  Week 240, HBsAg Seroconversion, n=77 | 1.3 [0.0 to 4.5]

12. Secondary Outcome: Percentage of Participants Who Experienced Viral Breakthrough
Description: Viral breakthrough was defined as >=1 log10 increase in HBV DNA from nadir determined by two sequential HBV DNA measurements. Percentage of Participants who experienced viral breakthrough at Week 48, Week 96, Week 144, Week 192 and Week 240 is presented.
Time Frame: Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 195
Percentage of Participants
  Week 48, n=195 | 0 [NA to NA] — NA indicates that 95% CI could not be calculated due to insufficient participants with events
  Week 96, n=195 | 0 [NA to NA] — NA indicates that 95% CI could not be calculated due to insufficient participants with events
  Week 144, n=185: number analyzed (Participants) | 185
  Week 144, n=185 | 0.5 [0.0 to 1.9]
  Week 192, n=180: number analyzed (Participants) | 180
  Week 192, n=180 | 1.1 [0.0 to 2.9]
  Week 240, n=161: number analyzed (Participants) | 161
  Week 240, n=161 | 0.6 [0.0 to 2.1]

13. Secondary Outcome: Percentage of Participants With Histological Improvement at Week 216
Description: The Knodell scoring system, also called the Histologic Activity Index (HAI), classifies liver biopsy specimens according to scores into 4 categories of histologic features: (I) Periportal or periseptal interface hepatitis (piecemeal necrosis) (scores from 0, 1, 2, 3, 4 or 10); (II) Confluent necrosis (scores from 0, 1, 3, 4, 5, 6 or 10); (III) Focal (spotty) lytic necrosis, apoptosis and focal inflammation (scores from 0, 1, 2, 3, 4 or 10); (IV) Portal inflammation (scores from 0, 1, 2, 3, 4 or 10). Histological improvement is considered as a reduction of two or more points in the Knodell necroinflammatory score with no increase in fibrosis.
Time Frame: Week 216
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 31
Percentage of participants | 45.2 [26.0 to 64.3]

14. Secondary Outcome: Percentage of Participants With Cirrhosis Reversal at Week 216
Description: Cirrhosis reversal was defined as a reduction of one or more points in the Ishak score with no evidence of cirrhosis. The Ishak liver fibrosis score ranges from 0 indicating no fibrosis to 6 indicating cirrhosis.
Time Frame: Week 216
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 31
Percentage of participants | 41.9 [23.0 to 60.9]

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and Non-serious TEAEs
Description: An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is defined as AE that occurred on or after the first dose date of study drug. SAE is any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, is a congenital anomaly/birth defect and other situations according to medical or scientific judgement or events possible drug-induced liver injury with hyperbilirubinemia.
Time Frame: Up to Week 240
Population: Safety Analysis Population was defined as all participants who received at least one dose of study medication and have at least one post Baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 195
Participants
  Any TEAEs | 139
  Serious TEAE | 34
  Non-serious TEAE | 129

16. Secondary Outcome: Change From Baseline in Hematology Parameters: White Blood Cells (WBC), Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, WBC, lymphocytes, monocytes, neutrophils and platelets. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Week 48, Week 96, Week 144, Week 192 and Week 240
Population: Safety analysis Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 191
10^9 cells per liter
  Week 48, WBC, n=191 | 0.02 (1.264)
  Week 96, WBC, n=188: number analyzed (Participants) | 188
  Week 96, WBC, n=188 | 0.09 (1.380)
  Week 144, WBC, n=185: number analyzed (Participants) | 185
  Week 144, WBC, n=185 | -0.12 (1.378)
  Week 192, WBC, n=179: number analyzed (Participants) | 179
  Week 192, WBC, n=179 | 0.12 (1.412)
  Week 240, WBC, n=160: number analyzed (Participants) | 160
  Week 240, WBC, n=160 | 0.06 (1.434)
  Week 48, Neutrophils, n=191 | 0.08 (1.051)
  Week 96, Neutrophils, n=188: number analyzed (Participants) | 188
  Week 96, Neutrophils, n=188 | 0.21 (1.184)
  Week 144, Neutrophils, n=185: number analyzed (Participants) | 185
  Week 144, Neutrophils, n=185 | 0.07 (1.162)
  Week 192, Neutrophils, n=179: number analyzed (Participants) | 179
  Week 192, Neutrophils, n=179 | 0.26 (1.197)
  Week 240, Neutrophils, n=160: number analyzed (Participants) | 160
  Week 240, Neutrophils, n=160 | 0.28 (1.194)
  Week 48, Lymphocytes, n=191 | 0.00 (0.438)
  Week 96, Lymphocytes, n=188: number analyzed (Participants) | 188
  Week 96, Lymphocytes, n=188 | -0.06 (0.511)
  Week 144, Lymphocytes, n=185: number analyzed (Participants) | 185
  Week 144, Lymphocytes, n=185 | -0.13 (0.422)
  Week 192, Lymphocytes, n=179: number analyzed (Participants) | 179
  Week 192, Lymphocytes, n=179 | -0.10 (0.442)
  Week 240, Lymphocytes, n=160: number analyzed (Participants) | 160
  Week 240, Lymphocytes, n=160 | -0.15 (0.483)
  Week 48, Monocytes, n=191 | -0.032 (0.1056)
  Week 96, Monocytes, n=188: number analyzed (Participants) | 188
  Week 96, Monocytes, n=188 | -0.033 (0.1113)
  Week 144, Monocytes, n=185: number analyzed (Participants) | 185
  Week 144, Monocytes, n=185 | -0.035 (0.1244)
  Week 192, Monocytes, n=179: number analyzed (Participants) | 179
  Week 192, Monocytes, n=179 | -0.025 (0.1162)
  Week 240, Monocytes, n=160: number analyzed (Participants) | 160
  Week 240, Monocytes, n=160 | -0.005 (0.1664)
  Week 48, Eosinophils, n=191 | -0.02 (0.114)
  Week 96, Eosinophils, n=188: number analyzed (Participants) | 188
  Week 96, Eosinophils, n=188 | -0.02 (0.164)
  Week 144, Eosinophils, n=185: number analyzed (Participants) | 185
  Week 144, Eosinophils, n=185 | -0.04 (0.237)
  Week 192, Eosinophils, n=179: number analyzed (Participants) | 179
  Week 192, Eosinophils, n=179 | -0.03 (0.248)
  Week 240, Eosinophils, n=160: number analyzed (Participants) | 160
  Week 240, Eosinophils, n=160 | -0.03 (0.251)
  Week 48, Basophils, n=191 | 0.00 (0.017)
  Week 96, Basophils, n=188: number analyzed (Participants) | 188
  Week 96, Basophils, n=188 | 0.00 (0.019)
  Week 144, Basophils, n=184: number analyzed (Participants) | 184
  Week 144, Basophils, n=184 | 0.01 (0.025)
  Week 192, Basophils, n=179: number analyzed (Participants) | 179
  Week 192, Basophils, n=179 | 0.01 (0.021)
  Week 240, Basophils, n=160: number analyzed (Participants) | 160
  Week 240, Basophils, n=160 | 0.01 (0.033)
  Week 48, Platelets, n=191 | 7.8 (31.45)
  Week 96, Platelets, n=188: number analyzed (Participants) | 188
  Week 96, Platelets, n=188 | 14.1 (32.46)
  Week 144, Platelets, n=185: number analyzed (Participants) | 185
  Week 144, Platelets, n=185 | 20.6 (42.02)
  Week 192, Platelets, n=179: number analyzed (Participants) | 179
  Week 192, Platelets, n=179 | 25.7 (42.56)
  Week 240, Platelets, n=160: number analyzed (Participants) | 160
  Week 240, Platelets, n=160 | 26.6 (38.39)

17. Secondary Outcome: Change From Baseline in Hemoglobin (Hb)
Description: Blood samples were collected to analyze Hb values. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 191
Grams per liter
  Week 48, n=191 | -0.6 (10.12)
  Week 96, n=188: number analyzed (Participants) | 188
  Week 96, n=188 | 0.2 (11.63)
  Week 144, n=185: number analyzed (Participants) | 185
  Week 144, n=185 | 0.9 (11.26)
  Week 192, n=179: number analyzed (Participants) | 179
  Week 192, n=179 | -0.3 (12.61)
  Week 240, n=160: number analyzed (Participants) | 160
  Week 240, n=160 | 1.2 (12.71)

18. Secondary Outcome: Change From Baseline in Red Blood Cells (RBC)
Description: Blood samples were collected to analyze RBC values. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 191
Trillion cells per liter
  Week 48, n=191 | 0.11 (0.306)
  Week 96, n=188: number analyzed (Participants) | 188
  Week 96, n=188 | 0.13 (0.344)
  Week 144, n=185: number analyzed (Participants) | 185
  Week 144, n=185 | 0.15 (0.340)
  Week 192, n=179: number analyzed (Participants) | 179
  Week 192, n=179 | 0.10 (0.363)
  Week 240, n=160: number analyzed (Participants) | 160
  Week 240, n=160 | 0.12 (0.341)

19. Secondary Outcome: Change From Baseline in Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma-Glutamyltransferase (GGT), Creatinine Phosphokinase (CK), Lactose Dehydrogenase (LDH)
Description: Blood samples were collected to analyze the chemistry parameters: ALT, ALP, AST, GGT, CK, LDH. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 191
Units per liter
  Week 48, ALT, n=190: number analyzed (Participants) | 190
  Week 48, ALT, n=190 | -23.98 (59.452)
  Week 96, ALT, n=187: number analyzed (Participants) | 187
  Week 96, ALT, n=187 | -28.99 (56.983)
  Week 144, ALT, n=185: number analyzed (Participants) | 185
  Week 144, ALT, n=185 | -28.99 (56.983)
  Week 192, ALT, n=178: number analyzed (Participants) | 178
  Week 192, ALT, n=178 | -31.79 (57.955)
  Week 240, ALT, n=158: number analyzed (Participants) | 158
  Week 240, ALT, n=158 | -32.02 (63.157)
  Week 48, AST, n=191 | -14.69 (36.674)
  Week 96, AST, n=188: number analyzed (Participants) | 188
  Week 96, AST, n=188 | -17.97 (36.057)
  Week 144, AST, n=184: number analyzed (Participants) | 184
  Week 144, AST, n=184 | -18.10 (36.809)
  Week 192, AST, n=178: number analyzed (Participants) | 178
  Week 192, AST, n=178 | -19.82 (36.312)
  Week 240, AST, n=158: number analyzed (Participants) | 158
  Week 240, AST, n=158 | -20.24 (43.908)
  Week 48, ALP, n=190: number analyzed (Participants) | 190
  Week 48, ALP, n=190 | 10.18 (20.288)
  Week 96, ALP, n=188: number analyzed (Participants) | 188
  Week 96, ALP, n=188 | 2.60 (28.233)
  Week 144, ALP, n=185: number analyzed (Participants) | 185
  Week 144, ALP, n=185 | -2.20 (26.555)
  Week 192, ALP, n=177: number analyzed (Participants) | 177
  Week 192, ALP, n=177 | -0.94 (31.604)
  Week 240, ALP, n=158: number analyzed (Participants) | 158
  Week 240, ALP, n=158 | -4.68 (27.596)
  Week 48, GGT, n=190: number analyzed (Participants) | 190
  Week 48, GGT, n=190 | -17.88 (32.753)
  Week 96, GGT, n=188: number analyzed (Participants) | 188
  Week 96, GGT, n=188 | -22.20 (34.866)
  Week 144, GGT, n=185: number analyzed (Participants) | 185
  Week 144, GGT, n=185 | -24.69 (39.764)
  Week 192, GGT, n=175: number analyzed (Participants) | 175
  Week 192, GGT, n=175 | -24.07 (38.609)
  Week 240, GGT, n=152: number analyzed (Participants) | 152
  Week 240, GGT, n=152 | -27.26 (42.932)
  Week 48 CK, n=188: number analyzed (Participants) | 188
  Week 48 CK, n=188 | 10.51 (103.515)
  Week 96, CK, n=185: number analyzed (Participants) | 185
  Week 96, CK, n=185 | 16.77 (141.961)
  Week 144, CK, n=182: number analyzed (Participants) | 182
  Week 144, CK, n=182 | 5.96 (101.897)
  Week 192, CK, n=173: number analyzed (Participants) | 173
  Week 192, CK, n=173 | 13.72 (106.986)
  Week 240, CK, n=156: number analyzed (Participants) | 156
  Week 240, CK, n=156 | 2.79 (105.349)
  Week 48, LDH, n=187: number analyzed (Participants) | 187
  Week 48, LDH, n=187 | -10.62 (52.851)
  Week 96, LDH, n=185: number analyzed (Participants) | 185
  Week 96, LDH, n=185 | -10.21 (48.112)
  Week 144, LDH, n=180: number analyzed (Participants) | 180
  Week 144, LDH, n=180 | 3.34 (73.047)
  Week 192, LDH, n=172: number analyzed (Participants) | 172
  Week 192, LDH, n=172 | -18.45 (87.931)
  Week 240, LDH, n=155: number analyzed (Participants) | 155
  Week 240, LDH, n=155 | 25.79 (87.464)

20. Secondary Outcome: Change From Baseline in Chemistry Parameters: Total Bilirubin, Direct Bilirubin, Serum Creatinine
Description: Blood samples were collected to analyze the chemistry parameters: total billirubin,direct bilirubin and serum creatinine. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 191
Micromoles per liter
  Week 48, total bilirubin, n=191 | -1.485 (7.1347)
  Week 96, total bilirubin, n=188: number analyzed (Participants) | 188
  Week 96, total bilirubin, n=188 | -1.823 (6.7167)
  Week 144, total bilirubin, n=185: number analyzed (Participants) | 185
  Week 144, total bilirubin, n=185 | -2.665 (7.1281)
  Week 192, total bilirubin, n=177: number analyzed (Participants) | 177
  Week 192, total bilirubin, n=177 | -2.791 (6.9230)
  Week 240, total bilirubin, n=158: number analyzed (Participants) | 158
  Week 240, total bilirubin, n=158 | -1.772 (6.9786)
  Week 48, direct bilirubin, n=191 | -0.296 (3.1229)
  Week 96, direct bilirubin, n=188: number analyzed (Participants) | 188
  Week 96, direct bilirubin, n=188 | -0.462 (3.1875)
  Week 144, direct bilirubin, n=185: number analyzed (Participants) | 185
  Week 144, direct bilirubin, n=185 | -0.713 (3.4898)
  Week 192, direct bilirubin, n=178: number analyzed (Participants) | 178
  Week 192, direct bilirubin, n=178 | -0.780 (3.5942)
  Week 240, direct bilirubin, n=157: number analyzed (Participants) | 157
  Week 240, direct bilirubin, n=157 | -0.599 (3.5608)
  Week 48, serum creatinine, n=191 | 1.03 (7.020)
  Week 96, serum creatinine, n=188: number analyzed (Participants) | 188
  Week 96, serum creatinine, n=188 | 1.10 (7.597)
  Week 144, serum creatinine, n=184: number analyzed (Participants) | 184
  Week 144, serum creatinine, n=184 | 0.76 (9.122)
  Week 192, serum creatinine, n=178: number analyzed (Participants) | 178
  Week 192, serum creatinine, n=178 | 1.37 (8.591)
  Week 240, serum creatinine, n=159: number analyzed (Participants) | 159
  Week 240, serum creatinine, n=159 | 1.35 (9.879)

21. Secondary Outcome: Change From Baseline in Chemistry Parameters: Albumin and Total Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin and total protein. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 191
Grams per liter
  Week 48, albumin, n=191 | 1.06 (3.063)
  Week 96, albumin, n=188: number analyzed (Participants) | 188
  Week 96, albumin, n=188 | 1.23 (3.313)
  Week 144, albumin, n=185: number analyzed (Participants) | 185
  Week 144, albumin, n=185 | 1.86 (3.675)
  Week 192, albumin, n=175: number analyzed (Participants) | 175
  Week 192, albumin, n=175 | 1.65 (3.780)
  Week 240, albumin, n=158: number analyzed (Participants) | 158
  Week 240, albumin, n=158 | 1.81 (3.790)
  Week 48, total protein, n=191 | -1.01 (5.273)
  Week 96, total protein, n=188: number analyzed (Participants) | 188
  Week 96, total protein, n=188 | -0.21 (5.397)
  Week 144, total protein, n=185: number analyzed (Participants) | 185
  Week 144, total protein, n=185 | 0.27 (5.065)
  Week 192, total protein, n=175: number analyzed (Participants) | 175
  Week 192, total protein, n=175 | -0.94 (5.175)
  Week 240, total protein, n=158: number analyzed (Participants) | 158
  Week 240, total protein, n=158 | -1.61 (5.829)

22. Secondary Outcome: Change From Baseline in Chemistry Parameter: Blood Urea Nitrogen (BUN), Potassium, Sodium, Chloridion, Phosphorus, Calcium and Fasting Blood Glucose
Description: Blood samples were collected to analyze the chemistry parameters: BUN, potassium, sodium, chloridion, phosphorus,calcium and fasting blood glucose. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 191
Millimoles per liter
  Week 48, BUN, n=191 | -0.046 (1.1067)
  Week 96, BUN, n=188: number analyzed (Participants) | 188
  Week 96, BUN, n=188 | 0.000 (1.1875)
  Week 144, BUN, n=184: number analyzed (Participants) | 184
  Week 144, BUN, n=184 | 0.037 (1.0892)
  Week 192, BUN, n=178: number analyzed (Participants) | 178
  Week 192, BUN, n=178 | 0.143 (1.1234)
  Week 240, BUN, n=155: number analyzed (Participants) | 155
  Week 240, BUN, n=155 | 0.131 (1.1358)
  Week 48, Potassium, n=191 | -0.001 (0.3703)
  Week 96, Potassium, n=186: number analyzed (Participants) | 186
  Week 96, Potassium, n=186 | 0.002 (0.3230)
  Week 144, Potassium, n=184: number analyzed (Participants) | 184
  Week 144, Potassium, n=184 | -0.039 (0.3871)
  Week 192, Potassium, n=178: number analyzed (Participants) | 178
  Week 192, Potassium, n=178 | 0.015 (0.4223)
  Week 240, Potassium, n=158: number analyzed (Participants) | 158
  Week 240, Potassium, n=158 | -0.013 (0.3946)
  Week 48, Sodium, n=191 | 0.21 (3.495)
  Week 96, Sodium, n=186: number analyzed (Participants) | 186
  Week 96, Sodium, n=186 | -0.02 (3.121)
  Week 144, Sodium, n=184: number analyzed (Participants) | 184
  Week 144, Sodium, n=184 | 0.35 (2.730)
  Week 192, Sodium, n=178: number analyzed (Participants) | 178
  Week 192, Sodium, n=178 | 0.38 (2.998)
  Week 240, Sodium, n=158: number analyzed (Participants) | 158
  Week 240, Sodium, n=158 | -0.13 (2.707)
  Week 48, Chloridion, n=191 | -0.13 (3.600)
  Week 96, Chloridion, n=186: number analyzed (Participants) | 186
  Week 96, Chloridion, n=186 | 0.40 (3.535)
  Week 144, Chloridion, n=183: number analyzed (Participants) | 183
  Week 144, Chloridion, n=183 | 0.35 (3.492)
  Week 192, Chloridion, n=178: number analyzed (Participants) | 178
  Week 192, Chloridion, n=178 | 0.77 (3.142)
  Week 240, Chloridion, n=158: number analyzed (Participants) | 158
  Week 240, Chloridion, n=158 | 0.49 (3.364)
  Week 48, Phosphorus, n=190: number analyzed (Participants) | 190
  Week 48, Phosphorus, n=190 | -0.044 (0.1724)
  Week 96, Phosphorus, n=187: number analyzed (Participants) | 187
  Week 96, Phosphorus, n=187 | -0.038 (0.1632)
  Week 144, Phosphorus, n=184: number analyzed (Participants) | 184
  Week 144, Phosphorus, n=184 | -0.037 (0.1955)
  Week 192, Phosphorus, n=175: number analyzed (Participants) | 175
  Week 192, Phosphorus, n=175 | -0.059 (0.1876)
  Week 240, Phosphorus, n=159: number analyzed (Participants) | 159
  Week 240, Phosphorus, n=159 | -0.042 (0.2009)
  Week 48, Calcium, n=190: number analyzed (Participants) | 190
  Week 48, Calcium, n=190 | -0.023 (0.1513)
  Week 96, Calcium, n=187: number analyzed (Participants) | 187
  Week 96, Calcium, n=187 | -0.006 (0.1652)
  Week 144, Calcium, n=184: number analyzed (Participants) | 184
  Week 144, Calcium, n=184 | -0.022 (0.1605)
  Week 192, Calcium, n=178: number analyzed (Participants) | 178
  Week 192, Calcium, n=178 | -0.004 (0.1470)
  Week 240, Calcium, n=158: number analyzed (Participants) | 158
  Week 240, Calcium, n=158 | -0.006 (0.1558)
  Week 48, Fasting Blood Glucose, n=191 | -0.162 (0.7154)
  Week 96, Fasting Blood Glucose, n=188: number analyzed (Participants) | 188
  Week 96, Fasting Blood Glucose, n=188 | -0.109 (0.7139)
  Week 144, Fasting Blood Glucose, n=185: number analyzed (Participants) | 185
  Week 144, Fasting Blood Glucose, n=185 | -0.094 (0.8979)
  Week 192, Fasting Blood Glucose, n=177: number analyzed (Participants) | 177
  Week 192, Fasting Blood Glucose, n=177 | -0.052 (0.7548)
  Week 240, Fasting Blood Glucose, n=158: number analyzed (Participants) | 158
  Week 240, Fasting Blood Glucose, n=158 | 0.052 (1.2197)

23. Secondary Outcome: Change From Baseline in Chemistry Parameters: Creatinine Clearance Rate
Description: Blood samples were collected to analyze the chemistry parameters: creatinine clearance rate. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Milliliter per minute (mL/min)
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 190
Milliliter per minute (mL/min)
  Week 48, n=190 | -3.064 (11.5995)
  Week 96, n=188: number analyzed (Participants) | 188
  Week 96, n=188 | -4.214 (12.7883)
  Week 144, n=184: number analyzed (Participants) | 184
  Week 144, n=184 | -4.324 (15.3937)
  Week 192, n=177: number analyzed (Participants) | 177
  Week 192, n=177 | -6.599 (13.8858)
  Week 240, n=155: number analyzed (Participants) | 155
  Week 240, n=155 | -6.658 (16.5351)

24. Secondary Outcome: Change From Baseline in Chemistry Parameters: Estimated Glomerular Filtration Rate (eGFR)
Description: Blood samples were collected to analyze the chemistry parameters: eGFR. Day 0 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 0) and at Week 48, Week 96, Week 144, Week 192 and Week 240
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mL/minute per 1.73 square meter
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
Number analyzed (Participants) | 191
mL/minute per 1.73 square meter
  Week 48, n=191 | -0.86 (6.581)
  Week 96, n=188: number analyzed (Participants) | 188
  Week 96, n=188 | -0.87 (7.078)
  Week 144, n=185: number analyzed (Participants) | 185
  Week 144, n=185 | -0.68 (8.368)
  Week 192, n=180: number analyzed (Participants) | 180
  Week 192, n=180 | -1.06 (8.442)
  Week 240, n=161: number analyzed (Participants) | 161
  Week 240, n=161 | -1.42 (9.609)

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious TEAEs and serious TEAEs were collected up to 240 weeks from the start of the treatment.
Description: Safety analysis population was used to collect the adverse events
Arm/Group | Tenofovir Disoproxil Fumarate 300 mg
All-Cause Mortality (participants affected / at risk) | 2/195
Serious Adverse Events (participants affected / at risk) | 34/195
Other Adverse Events (participants affected / at risk) | 129/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir Disoproxil Fumarate 300 mg (N=195)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Rheumatic fever (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Uterine adhesions (Reproductive system and breast disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Hypersplenism (Blood and lymphatic system disorders) | 1
Rheumatic heart disease (Cardiac disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Chest X-ray abnormal (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir Disoproxil Fumarate 300 mg (N=195)
Upper respiratory tract infection (Infections and infestations) | 36
Urinary tract infection (Infections and infestations) | 11
Nasopharyngitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Pulmonary tuberculosis (Infections and infestations) | 2
Urethritis (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Myringitis (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Tonsillitis bacterial (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Ascites (Gastrointestinal disorders) | 6
Toothache (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Epigastric discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Chronic gastritis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Abdominal mass (Gastrointestinal disorders) | 1
Dysbacteriosis (Gastrointestinal disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Blood creatine phosphokinase increased (Investigations) | 9
Protein urine present (Investigations) | 4
Blood phosphorus decreased (Investigations) | 3
Alpha 1 foetoprotein increased (Investigations) | 3
Blood urine present (Investigations) | 2
Weight decreased (Investigations) | 2
Blood uric acid increased (Investigations) | 2
Blood glucose increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Red blood cells urine positive (Investigations) | 1
Platelet count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Hepatitis B DNA increased (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Creatinine renal clearance decreased (Investigations) | 1
Blood urine (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 9
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Splenomegaly (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 5
Hepatic pain (Hepatobiliary disorders) | 2
Liver injury (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 2
Hepatic steatosis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Gallbladder polyp (Hepatobiliary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Renal injury (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Animal bite (Injury, poisoning and procedural complications) | 2
Ligament sprain (Injury, poisoning and procedural complications) | 2
Joint injury (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Skin wound (Injury, poisoning and procedural complications) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Leukoderma (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 2
Uterine enlargement (Reproductive system and breast disorders) | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 1
Breast hyperplasia (Reproductive system and breast disorders) | 1
Menstruation delayed (Reproductive system and breast disorders) | 1
Hypertension (Vascular disorders) | 5
Pyrexia (General disorders) | 1
Fatigue (General disorders) | 1
Chest pain (General disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vitreous floaters (Eye disorders) | 1
Retinal vein occlusion (Eye disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Bradycardia (Cardiac disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Transaminases increased (Investigations) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT02224456/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT02224456/SAP_001.pdf